CLINICAL TRIAL: NCT00951392
Title: Implication of Metabolic and Genomic Modifications in Elderly Subjects
Acronym: COMPALICLAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Martine Laville PhD, MD, Hospices Civils de Lyon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008.547
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2010-03

CONDITIONS: Insulin Sensitivity; Aging
Keywords: Insulin sensitivity; aging; lipid metabolism; hyperinsulinemic clamp; gene expression; sirtuins
MeSH Terms: conditions — Insulin Resistance | interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problematic aging (Experimental)
  Interventions: Drug: euglycemic hyperinsulinemic clamp; Procedure: muscle biopsy; Device: indirect calorimetry
- successful aging (Experimental)
  Interventions: Drug: euglycemic hyperinsulinemic clamp; Procedure: muscle biopsy; Device: indirect calorimetry

INTERVENTIONS:
Drug: euglycemic hyperinsulinemic clamp — Insulin perfusion at 1 mU.kg-1.min-1
  Glucose perfusion to maintain euglycemia at 5,0 ± 0,5 mmol/l
  Blood tests
Procedure: muscle biopsy — Gene expression in muscle tissue will be studied with two approaches :
  * Candidate gene approach by quantitative RT-PCR : genes involved in the carbohydrates and lipids metabolism including lipid oxidation in muscle (lipid carriers, PPARs), expression of 7 sirtuins isoforms as well as some of their target genes (NFkB, PGC1a)
  * Global transcriptome analysis by DNA Chip
Device: indirect calorimetry — energy expenditure measurement

SUMMARY:
An increase of longevity and of the number of men and women older than 60 years old is observed in most industrialized countries. Aging is a complex, multifactorial and continuous process involving physical and biological modifications such as a notably decrease in glucose tolerance and type 2 diabetes risk. Insulin sensitivity follow-up during aging is difficult mainly because of many confounding factors (environment, lifestyle).

In 2006, SUVIMAX 2 study began, based on the monitoring of volunteers who participated in former SUVIMAX study (1994-2003). This study was a randomised trial which was designed to study the link between a low antioxidant intake and risk of cancer or ischemic heart disease. The subjects recently had a health check-up including complete information about their diet, physical and neurosensory status. Based on these data, a score was established to classify subjects according to their quality of aging ("successful aging versus "problematic aging") These volunteers, who undertook a 13-year follow-up (dietary and medical status), constitute the reference population to determine the mechanisms involved in the insulin resistance development in aging.

The purpose of our research work is to determine whether the quality of aging could influence insulin sensitivity, by studying metabolic profile and change in gene expression (genes involved in glucose metabolism and metabolic senescence in muscle tissue) during aging.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers from the cohort aging SUVIMAX 2
* Men and Women
* over 60 years
* BMI between 18 and 35 kg/m2 (including terminals)
* Normal medical check up
* Blood pressure < 140/90 mmHg
* Normal glycemia, lipid profile
* sedentary or moderate physical activity (maximum 4 hours per week)

Exclusion Criteria:

* Biological results or anormal chek-up
* medical or surgical history not compatible with study
* severe digestive, cardiovascular, renal, liver or tumor disorders history in the 5 last years
* infectious or inflammatory disease within 2 months
* surgical history within 3 months
* bood donation within 2 months
* coagulation disease, anticoagulant or antiplatelet agents (aspirin ...) treatment
* xylocaïn allergy
* claustrophobia
* Drug that could affect insulin sensitivity (beta blockers, lipid lowering, oral antidiabetics, insulin, , steroids)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Comparison of metabolic profile (lipid metabolism and energy expenditure) and insulin sensitivity based on the aging quality | 120 minutes

SECONDARY OUTCOMES:
Gene expression in muscle tissue by quantitative RT-PCR: genes involved in the carbohydrates and lipids metabolism (lipid carriers, PPARs), 7 sirtuins isoforms and of their target genes (NFkB, PGC1a) | one day
Gene expression in muscle tissue by Global transcriptome analysis by DNA Chip | one day

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, MD, PhD, Principal Investigator — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de recherche en nutrition humaine Rhône-Alpes, Pierre-Bénite, France

REFERENCES:
- [Result] Betry C, Meugnier E, Pflieger M, Grenet G, Hercberg S, Galan P, Kesse-Guyot E, Vidal H, Laville M. High expression of CPT1b in skeletal muscle in metabolically healthy older subjects. Diabetes Metab. 2019 Apr;45(2):152-159. doi: 10.1016/j.diabet.2018.01.018. Epub 2018 Feb 12. PMID 29657112